CLINICAL TRIAL: NCT06535282
Title: The Brain Network Mechanism and Outcome After Surgical Intervention of Conductive Hearing Loss Accompanied by Tinnitus.
Brief Title: Brain Mechanism and Outcome of Surgical Intervention of Conductive Hearing Loss.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-328-01
Record Dates: First submitted 2024-05-22; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Conductive Hearing Loss; Tinnitus; Surgery
Keywords: Conductive Hearing Loss; tinnitus; surgery; outcome; EEG; mechanism
MeSH Terms: conditions — Hearing Loss, Conductive; Tinnitus | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- baseline (No Intervention): pre-operative period test results
- follow-up (Other): post-operative period test results
  Interventions: Other: surgery

INTERVENTIONS:
Other: surgery — Surgical treatment of conductive hearing loss with tinnitus
  Arms: follow-up

SUMMARY:
This study explores the brain region activation and remodeling of poor connections of brain regions in the postoperative outcomes of conductive hearing loss patients with tinnitus by comparing pre - and post-operative audiological assessment, tinnitus assessment and EEG data.

DETAILED DESCRIPTION:
This study explores the brain region activation and remodeling of poor connections of brain regions in the postoperative outcomes of conductive hearing loss patients with tinnitus by comparing pre - and post-operative audiological assessment, tinnitus assessment and EEG data. Including audiological assessment (pure tone audiometry, speech test), tinnitus assessment (tinnitus matching, tinnitus handicap inventory, tinnitus function index, visual analogue scale)and non-invasive brain imaging assessment (EEG, fNIRS).

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 60 years;
* diagnosed with conductive hearing loss with tinnitus;
* treated with surgery;
* able to cooperate with all Chinese version evaluation;
* right-handed.

Exclusion Criteria:

* Pure tone audiometry indicates that the average pure tone hearing threshold (500Hz, 1kHz, 2kHz, 4kHz) is > 91dB HL;
* acoustic neuroma, nasopharyngeal carcinoma;
* hearing loss caused by noise or drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
pure tone audiometry | 3-7 days before surgery, 1-12 months after surgery
  The air- conducted threshold, bone-conducted threshold and air- bone gap of each frequency of pure tone audiometry were used to compare pre - and post-operative hearing level.
speech test | 3-7 days before surgery, 1-12 months after surgery
  Speech audiometry was mainly used to analyze the speech recognition rate of patients before and after surgery
EEG activation | 3-7 days before surgery, 1-12 months after surgery
  EEG signals were used to explore the activation of brain regions and remodeling of poor connections in the postoperative outcomes of conductive hearing loss patients accompanied by with tinnitus. Power spectral density calculation, traceability analysis, functional connection, microstate, clustering coefficient, feature path length, feature path intermediation, and isocompatibility coefficient were collected and then analyzed.
tinnitus handicap inventory scores | 3-7 days before surgery, 1-12 months after surgery
  The total score of the THI scale and the scores of the three subscales(functional, emotional, and catastrophic) were collected before and after surgery for data analysis.

SECONDARY OUTCOMES:
tinnitus function index scores | 3-7 days before surgery, 1-12 months after surgery
  The total score of the TFI scale were collected before and after surgery for data analysis.
visual analogue scale | 3-7 days before surgery, 1-12 months after surgery
  The total score of the VAS were collected before and after surgery for data analysis. VAS scale 0-10. A score of 0 means that tinnitus has no impact on daily life, and a score of 10 means that tinnitus has an intolerable, fatal level of impact on daily life.
fNIRS activation | 3-7 days before surgery, 1-12 months after surgery
  fNIRS signals were used to explore the activation of brain regions and remodeling of poor connections in the postoperative outcomes of conductive hearing loss patients accompanied by with tinnitus. Power spectral density calculation, traceability analysis, functional connection, microstate, clustering coefficient, feature path length, feature path intermediation, and isocompatibility coefficient were collected and then analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No